CLINICAL TRIAL: NCT05813054
Title: Randomized, Double-blind, Placebo-controlled Clinical Study to Evaluate the Anti-aging Efficacy of Dermial®
Brief Title: Clinical Study to Evaluate the Anti-aging Efficacy of Dermial®
Acronym: DermiAge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioiberica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PJ-00106
Record Dates: First submitted 2023-02-17; First posted 2023-04-14 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2023-03

CONDITIONS: Skin Aging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HA matrix ingredient (Experimental): 1 cap/day
  Interventions: Dietary Supplement: HA matrix ingredient
- Placebo (Placebo Comparator): 1 cap/day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: HA matrix ingredient — 1 capsule/day
  Arms: HA matrix ingredient
Dietary Supplement: Placebo — 1 capsule/day
  Arms: Placebo

SUMMARY:
Oral supplement with an HA matrix ingredient composed of HA (60-75%), sulfated GAGs (≥10%), including DS and CS, and collagen (≥ 5%) to evaluate the hydration of the stratum corneum of facial skin in healthy women showing natural signs of age-related aging versus placebo

DETAILED DESCRIPTION:
This study includes 60 healthy volunteers in which will be evaluated if the oral supplement with Dermial [composed of HA (60-75%), sulfated GAGs (≥10%), including DS and CS, and collagen (≥ 5%)] is able to obtain differences versus placebo in healthy women showing natural signs of age-related aging versus placebo . It is a single-center, double-blind, randomized, placebo-controlled clinical study with proportion 1:1 between treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women between 35 and 65 years of age (inclusive), showing signs of physiological facial skin aging.
2. Women willing not to use any firming product, skin lightening, or any other topical or systemic medication known to affect skin aging or dyschromia during the study period.
3. Be informed of the nature of the study and give their IC in writing.
4. Women willing not to become pregnant during the course of the study, using contraceptive methods considered highly effective.

Exclusion Criteria:

1. Women with allergies to the ingredients in the investigational product.
2. Women who have used a dietary or nutricosmetic supplement containing HA, or who have undergone Botox or HA infiltrations, in the last 6 months prior to signing the IC.
3. Women who have undergone:

   * Superficial or medium-deep chemical peels or dermabrasion within the 6 weeks prior to signing the IC or inclusion document.
   * Deep facial chemical peel, non-ablative laser or fractional laser resurfacing in the 12 months prior to signing the IC or inclusion document.
   * Facial plastic surgery or a laser ablative procedure for photoaging in the 12 months prior to signing the IC or inclusion document.
4. Suspected uncontrolled disease, such as diabetes mellitus (DM), arterial hypertension (HT), hyperthyroidism or hypothyroidism, renal failure or liver failure.
5. Women who have received a PRP (Platelet Rich Plasma) injection as a treatment for aesthetic purposes, in the 3 months prior to inclusion by signing the IC.
6. Women who do not wish, for whatever reason, to take the supplements in the study.
7. Known pregnancy or lactation.
8. Presence of inflammatory skin disease such as psoriasis, atopic dermatitis, rosacea, acne or hidradenitis suppurativa.
9. Presence of active malignant pathologies or premalignant skin lesions such as actinic keratoses.
10. Psychiatric disorder that is not managed or any other circumstance or pathology that prevents the participant from understanding and/or complying with the study procedures.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Skin Moisture | Day 0, 12 week
  The changes in the hydration of the facial stratum corneum using the Corneometer® CM825 measuring device, range: 0-130 arbitrary units

SECONDARY OUTCOMES:
Skin Moisture | Day 0, 6 week, 12 week
  Evaluate changes in the hydration of the facial stratum corneum from baseline to 6 and 12 week by Corneometer® CM825 measuring device, range: 0-130 arbitrary units
Skin elasticity | Day 0, 6 week, 12 week
  The changes of skin elasticity by Cutometer ® Dual MPA 580 probe, range: 0-100%.
Skin hardness | Day 0, 6 week, 12 week
  The changes of Skin hardness by PCE-DDO 10 Durometer probe, range: 0-100 Shore O.
Skin Barrier | Day 0, 6 week, 12 week
  The changes of skin barrier in terms of TEWL (Trans Epidermal Water Loss) by Tewameter® TM300 probe, range: 0-80 (g*m-2*h-1).
Skin pH | Day 0, 6 week, 12 week
  The changes of skin pH by Skin-pH-Meter®PH905 probe, range: pH0 (acidic) - pH12 (alkaline).
Skin temperature | Day 0, 6 week, 12 week
  The changes of the skin temperature by Skin-Thermometer ST500 probe, range: 15°C-40°C.
Antioxidant capacity of the skin | Day 0, 6 week, 12 week
  The total antioxidant capacity will be measured in microcoulombs, using conductive hydrogel strips designed for the direct measurement of antioxidant capacity using eBQC®, range: 0-20 microcoulombs.
Erythema and skin melanin index | Day 0, 6 week, 12 week
  The erythema and melanin index will be measured in arbitrary units using the Mexameter® MX18 probe, range: 50-600 arbitrary units .
Skin stiffness/deformability | Day 0, 6 week, 12 week
  The changes of the stiffness/deformability by Indentometer IDM 800 probe, range: 0.00-3.00 millimeters.
Skin friction | Day 0, 6 week, 12 week
  The changes of the skin friction by Frictiometer FR-700, range: 0-30 arbitrary units .
Skin radiance | Day 0, 6 week, 12 week
  The changes of the skin radiance by Skin-Glossymeter GL 200 probe, range: 0-100 arbitrary units.
Facial Wrinkles and Fine lines of Crow's feet | Day 0, 6 week, 12 week
  Assessment of Reduction in Facial Wrinkles and Fine lines of Crow's feet area by VisioScan. It consists of a UV light camera and measures the skin surface profiles. (0-500 Rz)
Glogau Photodamage Scale | Day 0, 6 week, 12 week
  The change between the photodamage grade by dermatologist physical examination of treated area. The Glogau Photodamage Scale has a score from 1-4 (Type I: No wrinkles, Type II: Wrinkles in motion, Type III: Wrinkles at rest, Type IV: Only wrinkles), this scale represents a qualitative assessment to measure the severity of photodamage and wrinkles.
Satisfaction assessed | Day 0, 12 week
  Level of satisfaction with the sensation of skin hydration, texture, luminosity and smoothness using a self-administered 5-point Likert scale of intensity ( 1_Very dissatisfied; 2_Dissatisfied; 3_Neither satisfied nor dissatisfied; 4_Satisfied; 5_Very) satisfied
Safety assessment | Day 0 to 12 week (anytime)
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Arias, Principal Investigator — Hospital Virgen de las Nieves (Granada)
Locations (1):
- Hospital Virgen de las Nieves, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Montero-Vilchez T, Galvez-Martin P, Sanabria-de la Torre R, Cuenca-Barrales C, Molina-Leyva A, Martinez-Puig D, Velasco-Alvarez J, Arias-Santiago S. Oral Supplementation with a New Hyaluronic Acid Matrix Ingredient Improves Skin Brightness, Hydration, Smoothness, and Roughness: Results from a Randomized, Double-Blinded, Placebo-Controlled Study. Dermatol Ther (Heidelb). 2025 Aug;15(8):2099-2116. doi: 10.1007/s13555-025-01447-6. Epub 2025 Jun 11. PMID 40498387